CLINICAL TRIAL: NCT01263665
Title: Evaluation of the 25 Centimeter (cm) GORE® VIABAHN® Endoprosthesis With PROPATEN Bioactive Surface to Treat de Novo and/or Restenotic Lesions of the Superficial Femoral Artery (SFA)
Brief Title: Evaluation of the 25 Centimeter (cm) GORE® VIABAHN® Endoprosthesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VBL 10-04
Record Dates: First submitted 2010-12-08; First posted 2010-12-21 (Estimated); Results first posted 2014-02-24 (Estimated); Last update posted 2015-12-17 (Estimated); Status verified 2015-11

CONDITIONS: Peripheral Vascular Diseases
Keywords: stent-graft; superficial femoral artery; SFA; peripheral artery disease; PAD
MeSH Terms: conditions — Peripheral Vascular Diseases; Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 25cm Gore VIABAHN (Experimental): 25 cm GORE® VIABAHN® Endoprosthesis with PROPATEN Bioactive Surface
  Interventions: Device: 25 cm GORE® VIABAHN®

INTERVENTIONS:
Device: 25 cm GORE® VIABAHN® — 25 cm GORE® VIABAHN® Endoprosthesis with PROPATEN Bioactive Surface, possibly in conjunction with an additional overlapping VIABAHN® device (2.5, 5, 10, 15, or 25 cm lengths) based on the enrolled patient's lesion length (greater than or equal to 20 cm length).

SUMMARY:
The purpose of this study is to confirm the safety and performance of the 25 cm GORE® VIABAHN® Endoprosthesis with PROPATEN Bioactive Surface when used in the Superficial Femoral Artery.

ELIGIBILITY:
Inclusion Criteria:

* Lifestyle-limiting claudication or rest pain (meeting angiographic entry criteria) affecting a lower extremity (Rutherford Categories 2-4).
* A written informed consent form, which has been reviewed and approved by the Ethics Committee, has been read, understood and signed by the subject (or their legally authorized representative).
* At least 21 years of age.
* Noninvasive lower extremity arterial studies (ankle-brachial index, ABI) prior to (within 45 days) or at the time of the study procedure demonstrating a resting ankle-brachial index (ABI) ≤ 0.9 in the study limb. If ABI > 0.9, patient is eligible for study if toe-brachial index (TBI) is ≤ 0.5.
* A staged ipsilateral vascular procedure was not completed less than 30-days prior to the study procedure. Resting ABIs were completed prior to the study procedure a minimum of 30-days after the staged vascular procedure.
* Vascular treatment on the non-study leg for bilateral claudication was not performed less than 30-days prior to study procedure. Resting ABIs on the study limb were completed prior to the study procedure a minimum of 30-days after treatment on the non-study leg.
* Male, infertile female, or female of child bearing potential practicing an acceptable method of birth control with a negative pregnancy test within 7-days prior to study procedure.
* Projected life expectancy of greater than three years.
* The ability to comply with protocol follow-up requirements and required testing.
* Angiographic and Lesion Requirements (assessed intraoperatively):
* Lesion length of 20-35 cm located in the region beginning 1 cm below origin of the profunda femoris artery and ending 1 cm above the origin of the intercondylar fossa.
* De novo, post-percutaneous transluminal angioplasty (PTA), or post-atherectomy stenosis (> 50% at some point within the lesion by visual estimate) or occlusion of native SFA.
* Origin and proximal 1 cm of SFA are patent.
* Popliteal artery is patent from 1 cm above the origin of the intercondylar fossa distal to the radiographic knee joint.
* Reference vessel diameter of 4.0 - 7.5 mm in proximal and distal treatment segments within the SFA.
* Angiographic evidence of at least one patent tibial artery to the ankle that does not require intervention.
* Guidewire has successfully traversed lesion and is within the true lumen of the distal vessel.

Exclusion Criteria:

* Untreated flow-limiting aortoiliac occlusive disease.
* Any previous open surgical procedure in the target vessel or previous stent placement in the target vessel.
* Prior angioplasty on the target lesion performed less than 30 days prior to the study procedure (unless performed at time of the study procedure).
* Prior atherectomy on the target lesion performed less than 6 months prior to the study procedure (unless performed at time of the study procedure).
* Any previous treatment of the target vessel with a drug-eluting balloon.
* Femoral artery or popliteal artery aneurysm.
* Non-atherosclerotic disease resulting in occlusion (e.g. embolism, Buerger's disease, vasculitis).
* Tibial artery disease requiring treatment.
* Prior ipsilateral femoral artery bypass.
* Severe medical comorbidities (untreated coronary artery disease, congestive heart failure, severe chronic obstructive pulmonary disease, metastatic malignancy, dementia, etc.) or other medical condition that would preclude post-procedural ambulation.
* Popliteal artery vascular access at any time during procedure.
* Antegrade and retrograde vascular access on the same common femoral artery at the time of the SFA intervention.
* Major distal amputation (above the transmetatarsal) in the study or non-study limb.
* Septicemia.
* Any previously known coagulation disorder, including hypercoagulability.
* Morbid obesity or operative scarring that precludes percutaneous approach (physician's discretion).
* Contraindication to anticoagulation or antiplatelet therapy.
* Known allergies to stent/stent-graft components, including heparin sensitivity, allergy, or previous incidence of heparin-induced thrombocytopenia (HIT) type II.
* History of prior life-threatening reaction to contrast agent.
* Currently participating in another clinical research trial, unless approved by W. L. Gore & Associates in advance of study enrollment.
* Subject has one limb currently enrolled in the study.
* Current peritoneal or hemodialysis.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2010-12; Primary Completion 2012-08 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Zeller, Prof. Dr. med., Principal Investigator — Herzzentrum Bad Krozingen

REFERENCES:
- [Derived] Bohme T, Noory E, Brechtel K, Scheinert D, Bosiers M, Beschorner U, Zeller T. Heparin-Bonded Stent-Graft for the Treatment of TASC II C and D Femoropopliteal Lesions: 36-Month Results of the Viabahn 25 cm Trial. J Endovasc Ther. 2021 Apr;28(2):222-228. doi: 10.1177/1526602820965965. Epub 2020 Oct 12. PMID 33044119
- [Derived] Zeller T, Peeters P, Bosiers M, Lammer J, Brechtel K, Scheinert D, Rastan A, Noory E, Beschorner U. Heparin-bonded stent-graft for the treatment of TASC II C and D femoropopliteal lesions: the Viabahn-25 cm trial. J Endovasc Ther. 2014 Dec;21(6):765-74. doi: 10.1583/14-4790R.1. PMID 25453876

RESULTS

PARTICIPANT FLOW:
Groups:
- 25 cm Length GORE® VIABAHN® Endoprosthesis With PROPATEN Bioac: 25 cm length GORE® VIABAHN® Endoprosthesis with
  > PROPATEN Bioactive Surface Subjects
Period: Overall Study
Arm/Group | 25 cm Length GORE® VIABAHN® Endoprosthesis With PROPATEN Bioac
Started | 71
Completed | 62
Not Completed | 9
Not completed — Withdrew Consent | 1
Not completed — Lost to Follow-up | 3
Not completed — Death | 2
Not completed — Amputation above the ankle | 1
Not completed — Surgical Bypass | 2

BASELINE CHARACTERISTICS:
Population: Patients with de novo and/or restenotic lesions (post PTA) of the SFA, with a total lesion length of ≥ 20 cm based on visual estimate
Groups:
- Investigational Arm: 25 cm length GORE® VIABAHN® Endoprosthesis with> PROPATEN Bioactive Surface Subjects
Arm/Group | Investigational Arm
Number analyzed (Participants) | 71
Age, Continuous [Mean (Full Range); unit: years] | 66.7 [44.7 to 83.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 50
Region of Enrollment [Number; unit: participants]
  Austria | 3
  Germany | 51
  Belgium | 17

OUTCOME MEASURES:

1. Primary Outcome: Successful Completion of the Assigned Treatment
Description: Successful completion of the assigned treatment and postdeployment> stent length (of the first deployed 25 cm GORE> VIABAHN Endoprosthesis with PROPATEN Bioactive Surface)> being within 10% of pre-deployment stent length.
Time Frame: Evaluated immediately after the index procedure
Measure: Number; unit: percentage of subjects
Groups:
- 25 cm Length GORE® VIABAHN® Endoprosthesis With PROPATEN Bioac: 25 cm length GORE® VIABAHN® Endoprosthesis with> PROPATEN Bioactive Surface Subjects
Arm/Group | 25 cm Length GORE® VIABAHN® Endoprosthesis With PROPATEN Bioac
Number analyzed (Participants) | 71
percentage of subjects | 76.7

2. Primary Outcome: Device-related and Procedure-related Serious Adverse Events (SAEs) Within 30 Days of the Index Procedure
Time Frame: 30 Days post-procedure
Measure: Number; unit: participants
Arm/Group | 25 cm Length GORE® VIABAHN® Endoprosthesis With PROPATEN Bioac
Number analyzed (Participants) | 71
participants | 2

ADVERSE EVENTS:
Time Frame: Total through 2 years, data pulled as of 10Oct2014
Groups:
- 25 cm GORE VIABAHN: 25 cm GORE VIABAHN Endoprosthesis with PROPATEN Bioactive Surface
Arm/Group | 25 cm GORE VIABAHN
Serious Adverse Events (participants affected / at risk) | 39/71
Other Adverse Events (participants affected / at risk) | 20/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 25 cm GORE VIABAHN (N=71)
Acute coronary syndrome (Cardiac disorders) | 1
Angina pectoris (Cardiac disorders) | 3
Angina unstable (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 3
Coronary artery disease (Cardiac disorders) | 2
Coronary artery occlusion (Cardiac disorders) | 1
Impaired healing (General disorders) | 1
Inflammation (General disorders) | 3
Pyrexia (General disorders) | 1
Thrombosis in device (General disorders) | 17
Gangrene (Infections and infestations) | 1
Infection (Infections and infestations) | 3
Influenza (Infections and infestations) | 1
Arterial injury (Injury, poisoning and procedural complications) | 2
Contrast media reaction (Injury, poisoning and procedural complications) | 1
In-stent arterial restenosis (Injury, poisoning and procedural complications) | 9
C-reactive protein increased (Investigations) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Monoparesis (Nervous system disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2
Diabetic neuropathic ulcer (Skin and subcutaneous tissue disorders) | 1
Aortic aneurysm (Vascular disorders) | 1
Femoral arterial stenosis (Vascular disorders) | 10
Femoral artery occlusion (Vascular disorders) | 4
Intermittent claudication (Vascular disorders) | 2
Peripheral arterial occlusive disease (Vascular disorders) | 4
Peripheral ischaemia (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 25 cm GORE VIABAHN (N=71)
Oedema peripheral (General disorders) | 7
Vessel puncture site haematoma (General disorders) | 2
In-stent arterial restenosis (Injury, poisoning and procedural complications) | 16
C-reactive protein increased (Investigations) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5
Hypoaesthesia (Nervous system disorders) | 2
Ecchymosis (Skin and subcutaneous tissue disorders) | 2
Iliac artery stenosis (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Before the single-center publication is submitted or presented, the> Investigator will provide a copy to the Sponsor and allow the Sponsor 30 days to review and> comment. The Sponsor will review the publication for data accuracy only and not the> conclusions or interpretations. If the Sponsor requests, the publication will be delayed an> additional ninety (90) days, to allow Sponsor to ensure the protection of inventions or other> property of Sponsor.